CLINICAL TRIAL: NCT07024056
Title: Acute Acromioclavicular Joint Dislocation Rockwood Type (III&VI): Coracoclavicular Ligaments Reconstruction Associated With Acromioclavicular Ligament Reconstruction Versus Coracoclavicular Ligaments Reconstruction With Acromioclavicular Temporary k Wire Fixation
Brief Title: Acute ACJ Dislocation Type (III&VI): CC Ligaments Reconstruction With AC Ligament Reconstruction vs. CC Ligaments Reconstruction With AC Temporary k Wire Fixation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Amr Ahmed ElSherif, Resident, Shebin El-Kom Teaching Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACJ disruption management
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Acromioclavicular Joint; Acromioclavicular Joint Dislocation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- coracoclavicular ligaments reconstruction associated with acromioclavicular ligament reconstruction (Active Comparator): The Gracilis or SemiT graft will be harvested from the ipsilateral knee. The acromioclavicular joint will be exposed by the deltopectoral approach. A strap incision will be started from the acromioclavicular joint and extended distally towards the tip of coracoid process. 2 drill holes will be prepared on the superior cortex of the clavicle at the footprint of the original 2 ligaments, using a 4.5-mm drill bit. The 2 holes will be around 1.5 cm apart and the lateral hole was around 2 to 2.5 cm proximal to the distal end of the clavicle. Another 4.5 mm drill bit hole was created in the acromion. The graft exiting laterally around the coracoid is then passed through the conoid tunnel from inferior to superior and then passed through the acromial tunnel from superior to inferior to augment/reconstruct the AC joint capsule. The graft exiting the acromion tunnel is passed through the trapezoid tunnel from superior to inferior. The two free ends of the hamstring graft are tied together.
  Interventions: Procedure: coracoclavicular ligaments reconstruction associated with acromioclavicular ligament reconstruction
- coracoclavicular ligaments reconstruction with acromioclavicular temporary k wire fixation (Active Comparator): Two 2.4-mm tunnels corresponding to the origins of the conoid and trapezoid ligaments will be created through the distal clavicle, approximately 1.5cm apart from each other. The distal tunnel will be 2.5cm away from the AC joint. After harvesting the Gracilis or Semitendinosus from the ipsilateral leg, the graft was prepared with no. 2 Ethibond sutures and passed beneath the coracoid. Both ends of the graft will be passed inside out through the tunnels after enlarging the tunnels by 4.5 drill bit making a figure of 8 sling. The AC joint will be provisionally reduced with two 1.5/1.8-mm smooth K-wires while keeping the graft ends under adequate manual tension. The ends of the graft will be sutured onto themselves and the surrounding soft tissues.
  Interventions: Procedure: coracoclavicular ligaments reconstruction with acromioclavicular temporary k wire fixation

INTERVENTIONS:
Procedure: coracoclavicular ligaments reconstruction associated with acromioclavicular ligament reconstruction — The Gracilis or SemiT graft will be harvested from the ipsilateral knee. An oblique skin incision will be made starting from the ACJ and extended distally towards the tip of coracoid process. 2 drill holes will be prepared on the superior cortex of the clavicle at the footprint of the original 2 ligaments, using a 4.5-mm drill bit. The 2 holes will be around 1 cm apart and the lateral hole was around 2 to 2.5 cm proximal to the distal end of the clavicle. Another 4.5 mm drill bit hole was created in the acromion. The graft exiting laterally around the coracoid will be then passed through the conoid tunnel from inferior to superior and then passed through the acromial tunnel from superior to inferior. The graft exiting the acromion tunnel will be passed through the trapezoid tunnel from superior to inferior. The two free ends of the hamstring graft will be tied to one another with Ethibond No.2 sutures
  Arms: coracoclavicular ligaments reconstruction associated with acromioclavicular ligament reconstruction
Procedure: coracoclavicular ligaments reconstruction with acromioclavicular temporary k wire fixation — Two 2.4-mm tunnels corresponding to the origins of the conoid and trapezoid ligaments will be created through the distal clavicle, approximately 1.5cm apart from each other. The distal tunnel will be 2.5cm away from the AC joint. After harvesting the Gracilis or Semitendinosus from the ipsilateral leg, the graft was prepared with no. 2 Ethibond sutures and passed beneath the coracoid. Both ends of the graft will be passed inside out through the tunnels after enlarging the tunnels by 4.5 drill bit making a figure of 8 sling. The AC joint will be provisionally reduced with two 1.5/1.8-mm smooth K-wires while keeping the graft ends under adequate manual tension. The ends of the graft will be sutured onto themselves and the surrounding soft tissues. The wound will be closed in layers.
  Arms: coracoclavicular ligaments reconstruction with acromioclavicular temporary k wire fixation

SUMMARY:
The aim of this study is to compare the clinical and radiographical outcome of patients treated by coracoclavicular ligaments reconstruction associated with acromioclavicular ligament reconstruction versus coracoclavicular ligaments reconstruction acromioclavicular temporary k wire fixation in management of Acute AC dislocation Rockwood type (III&VI).

* Number of patients (20)
* Type of disease (AC dislocation Rockwood type (III&VI)
* follow up period (6 months)
* type of study: this is a clinical research study

DETAILED DESCRIPTION:
Acromioclavicular joint dislocation (ACD) is one of the most common shoulder injuries and is usually sports related. Acromioclavicular (AC) joint injuries account for about 12% of all shoulder injuries in clinical practice, a rate that increases to almost 40% in athletes participating in contact sports.

Epidemiological studies showed that most AC joint injuries occur in the third decade of life, and the gender distribution is 5:1 in favor of men. Acromioclavicular joint (ACJ) injuries have been reported to especially occur in 20- to 30-year-old male patients engaging in high-contact sports.

The mechanism of injury leading to AC joint dislocation can be direct or indirect. A direct force on the superior aspect of the acromion process, it happen due to fall onto the outer aspect of the shoulder, is the most common scenario. The acromioclavicular capsule-ligamentous structures fail with consecutive loading of the coraco-clavicular (CC) ligaments.

The Four components of the acromioclavicular (AC) capsular ligaments and the two components of the coracoclavicular (CC) ligaments contribute to AC joint stability depending upon the direction and magnitude of the force applied. The trapezoid ligament provides the major support against compressive loads applied along the axis of the clavicle and acts as a secondary restraint to superior translation. On the other hand, the conoid ligament contributes to both superior and anterior stability. Among the 4 AC capsular ligaments, the superior and posterior capsular ligaments, reinforced by the deltoid and trapezius muscle, are important due to their primary role in prevention of posterior translation. Despite the different contribution of each ligament on the stability of the AC joint, most current surgical techniques for complete AC joint dislocation focus on CC interval fixation to restore the CC ligaments.

Nonsurgical management is the mainstay of treatment for type I and II injuries, whereas surgery is usually recommended for type IV to VI injuries. The treatment for type III remains instead controversial as no clear treatment algorithm has been established.

Because of the distinct functional anatomy of the AC and CC ligaments, several studies provided good results focusing on anatomical surgical techniques that recreate those structures, rather than non-anatomical procedures that aim to improve function and stability regardless of restoration of anatomy of the torn ligaments. Although several anatomic reconstruction techniques are available, most of them showed promising results after conducting underpowered studies at short-term follow-up. Moreover, no gold standard has been identified yet.

Several surgical techniques have been described in the literature. Rockwood classified the early surgical treatments for AC joint instability into 4 groups: (1) AC ligament repairs, (2) CC ligaments repairs, (3) excision of the distal clavicle, and (4) dynamic muscle transfer. In addition, K-wires, screws, and plates have been used for temporary fixation of the AC joint. A better understanding of the anatomy and biomechanics of the AC joint and the coracoclavicular (CC) ligaments has led to advances in surgical techniques. Anatomic reconstructions using free grafts have become popular in recent years. In addition, arthroscopically assisted procedures using cortical fixation devices have become more popular.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years old.
* Acute AC dislocation Rockwood type VI.
* Acute AC dislocation Rockwood type III patients with pre-injury high level of activity (work or athletic activity).
* Patient is fit for surgery.
* Patient is willing to participate.

Exclusion Criteria:

* Chronic AC dislocation.
* AC dislocation Rockwood type (I, II, IV and VI).
* Previous surgery to the same shoulder, degenerative changes of the glenohumeral joint, shoulder infections, and concomitant neurologic diseases.
* Associated neurological disorders in the affected limb.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
complications | 12 months after surgery.
  Redislocations. Other local complications, eg. infection.

SECONDARY OUTCOMES:
Constant-Murley Score | 12 months after surgery.
  Constant-Murley Score (range: 0-100). Higher scores indicate better shoulder function. Scores above 80 generally reflect excellent shoulder performance.

REFERENCES:
- [Background] Frantz T, Ramkumar PN, Frangiamore S, Jones G, Soloff L, Kvit A, Curriero FC, Schickendantz M. Epidemiology of acromioclavicular joint injuries in professional baseball: analysis from the Major League Baseball Health and Injury Tracking System. J Shoulder Elbow Surg. 2021 Jan;30(1):127-133. doi: 10.1016/j.jse.2020.04.029. Epub 2020 Jun 9. PMID 32778383
- [Background] Saccomanno MF, Fodale M, Capasso L, Cazzato G, Milano G. Reconstruction of the coracoclavicular and acromioclavicular ligaments with semitendinosus tendon graft: a pilot study. Joints. 2014 May 8;2(1):6-14. eCollection 2014 Jan-Mar. PMID 25606535
- [Background] Pallis M, Cameron KL, Svoboda SJ, Owens BD. Epidemiology of acromioclavicular joint injury in young athletes. Am J Sports Med. 2012 Sep;40(9):2072-7. doi: 10.1177/0363546512450162. Epub 2012 Jun 15. PMID 22707749
- [Background] Sirin E, Aydin N, Mert Topkar O. Acromioclavicular joint injuries: diagnosis, classification and ligamentoplasty procedures. EFORT Open Rev. 2018 Jul 17;3(7):426-433. doi: 10.1302/2058-5241.3.170027. eCollection 2018 Jul. PMID 30233818
- [Background] Nolte PC, Lacheta L, Dekker TJ, Elrick BP, Millett PJ. Optimal Management of Acromioclavicular Dislocation: Current Perspectives. Orthop Res Rev. 2020 Mar 5;12:27-44. doi: 10.2147/ORR.S218991. eCollection 2020. PMID 32184680
- [Background] Shin SJ, Campbell S, Scott J, McGarry MH, Lee TQ. Simultaneous anatomic reconstruction of the acromioclavicular and coracoclavicular ligaments using a single tendon graft. Knee Surg Sports Traumatol Arthrosc. 2014 Sep;22(9):2216-22. doi: 10.1007/s00167-013-2569-x. Epub 2013 Jul 11. PMID 23842800
- [Background] Frank RM, Cotter EJ, Leroux TS, Romeo AA. Acromioclavicular Joint Injuries: Evidence-based Treatment. J Am Acad Orthop Surg. 2019 Sep 1;27(17):e775-e788. doi: 10.5435/JAAOS-D-17-00105. PMID 31008872
- [Background] Xara-Leite F, Andrade R, Moreira PS, Coutinho L, Ayeni OR, Sevivas N, Espregueira-Mendes J. Anatomic and non-anatomic reconstruction improves post-operative outcomes in chronic acromio-clavicular instability: a systematic review. Knee Surg Sports Traumatol Arthrosc. 2019 Dec;27(12):3779-3796. doi: 10.1007/s00167-019-05408-3. Epub 2019 Feb 26. PMID 30806755
- [Background] Moatshe G, Kruckeberg BM, Chahla J, Godin JA, Cinque ME, Provencher MT, LaPrade RF. Acromioclavicular and Coracoclavicular Ligament Reconstruction for Acromioclavicular Joint Instability: A Systematic Review of Clinical and Radiographic Outcomes. Arthroscopy. 2018 Jun;34(6):1979-1995.e8. doi: 10.1016/j.arthro.2018.01.016. Epub 2018 Mar 21. PMID 29573931
- [Background] Garofalo R, Ceccarelli E, Castagna A, Calvisi V, Flanagin B, Conti M, Krishnan SG. Open capsular and ligament reconstruction with semitendinosus hamstring autograft successfully controls superior and posterior translation for type V acromioclavicular joint dislocation. Knee Surg Sports Traumatol Arthrosc. 2017 Jul;25(7):1989-1994. doi: 10.1007/s00167-017-4509-7. Epub 2017 Apr 22. PMID 28434037